CLINICAL TRIAL: NCT05640258
Title: Seasickness Susceptability and Vestibular Time Constant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDF-1710-2016
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Seasickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- seasickness susceptibility and vestibular time constant (Experimental): All study participants underwent rotatory chair testing in a velocity step protocol to determine the Vestibular time constant.
  testing were preformed at baseline, before commencing active duty on a ship, 3 month and 6 month follow up after the beginning of active sailing.
  Interventions: Diagnostic Test: rotatory chair testing in a velocity step protocol.

INTERVENTIONS:
Diagnostic Test: rotatory chair testing in a velocity step protocol. — Tc was evaluated by the rotational velocity step test using the OtoaccessTM interface (Interacoustics Nydiag 200, Middlefart, Denmark). Subjects were seated on the rotatory chair wearing videonystagmography goggles with their heads supported and tilted 30° forward, thus bringing the horizontal semicircular canals plane perpendicular to the axis of rotation. Standard videonystagmography techniques were employed to record eye-movements. Subsequent to eye movements' calibration, the chair was accelerated about the yaw axis at 30°/sec2 to a maximal velocity of 90°/sec, followed by rotation at a constant velocity. After 57 seconds of constant velocity rotation, the chair was decelerated to zero velocity at 30°/sec2. The described velocity step was conducted both clockwise and counter-clockwise, giving a total run time of 4 minutes.

SUMMARY:
Participants were selected from the military navy crewmembers prior to commencing of active sailing.

A vestibular time constant was calculated based on velocity step testing on a rotatory chair at baseline, 3 months and 6 month following active sailing duty.

A seasickness questionnaire (WIKER) was completed during follow-up visits. study participants were divided to three groups based on WIKER score - susceptible , non-susceptible and habituating. Vestibular time constant was compared between study groups.

ELIGIBILITY:
Inclusion Criteria:

* healthy male Navy sailors in basic training

Exclusion Criteria:

* History of hearing loss
* Otoscopic findings of ear pathology
* An implanted electrode
* A finding of vestibulopathy upon otoneurological examination -
* Discontinuation of active sailing for any reason during study follow-up
* Withdrawal of informed consent.

Ages: 18 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
6 month follow up vestibular time constant measurement. | 6 months
  vestibular time constant in seconds is the measurement of decline in maximal slow phase velocity of eye movement during nystagmus to 37% of initial value produced by abrupt acceleration and declarations in a rotatory chair - step velocity protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli Naval Medical Institute, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
The data that supports the findings of this study are available upon request from the corresponding author, Tal D.

REFERENCES:
- [Derived] Lagami D, Gutkovich YE, Jamison A, Fonar Y, Tal D. Seasickness susceptibility and the vestibular time constant: a prospective study. Exp Brain Res. 2024 Jan;242(1):267-274. doi: 10.1007/s00221-023-06745-z. Epub 2023 Nov 28. PMID 38015244